CLINICAL TRIAL: NCT02452515
Title: A Single-blind, Multicenter Pilot Study to Investigate the Safety and Tolerability of a 14 Day Oral Treatment With Different Doses of the Chymase Inhibitor BAY1142524 in Comparison to Placebo in Clinically Stable Patients With Left-ventricular Dysfunction After Myocardial Infarction
Brief Title: A Single-blind Pilot Study to Investigate Safety and Tolerability of the Chymase Inhibitor BAY1142524 in Clinically Stable Patients With Left-ventricular Dysfunction
Acronym: CHIARA MIA 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 17055; 2014-005297-12 (EudraCT Number)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BAY1142524 (5 mg) (Experimental): 12 patients with left-ventricular dysfunction after myocardial infarction, 9 patients allocated to verum treatment, 3 patients allocated to placebo treatment
  Interventions: Drug: BAY1142524; Drug: Placebo
- BAY1142524 (10 mg) (Experimental): 12 patients with left-ventricular dysfunction after myocardial infarction, 9 patients allocated to verum treatment, 3 patients allocated to placebo treatment
  Interventions: Drug: BAY1142524; Drug: Placebo
- BAY1142524 (25 mg) (Experimental): 12 patients with left-ventricular dysfunction after myocardial infarction, 9 patients allocated to verum treatment, 3 patients allocated to placebo treatment
  Interventions: Drug: BAY1142524; Drug: Placebo
- BAY1142524 (50 mg) (Experimental): 12 patients with left-ventricular dysfunction after myocardial infarction, 9 patients allocated to verum treatment, 3 patients allocated to placebo treatment
  Interventions: Drug: BAY1142524; Drug: Placebo

INTERVENTIONS:
Drug: BAY1142524 — 5 mg BAY1142524 or placebo given as 5 mg IR tablet twice daily for 2 weeks
  Arms: BAY1142524 (5 mg)
Drug: BAY1142524 — 10 mg BAY1142524 or placebo given as 2 x 5 mg IR tablets twice daily as for 2 weeks
  Arms: BAY1142524 (10 mg)
Drug: BAY1142524 — 25 mg BAY1142524 or placebo given as 5 x 5 mg IR tablets twice daily for 2 weeks
  Arms: BAY1142524 (25 mg)
Drug: BAY1142524 — 50 mg BAY1142524 or placebo given 1 x 50 mg IR tablet once daily for 2 weeks
  Arms: BAY1142524 (50 mg)
Drug: Placebo — The patients will be treated orally with combinations of IR tablets containing placebo to achieve the indicated dosages.

SUMMARY:
The purpose of the trial is the analysis of safety and tolerability of the chymase inhibitor BAY1142524 in comparison to placebo using a 2 weeks treatment period in clinically stable patients with left-ventricular dysfunction after myocardial infarction. BAY1142524 or placebo will be given on top of evidence-based standard of care for left-ventricular dysfunction after myocardial infarction. Primary objectives are the analysis of safety and tolerability as evidenced by the incidence and severity of adverse events. BAY1142524 will be administered in a parallel group design using four doses (5, 10, 25 mg twice daily, and 50 mg once daily). Each dose group consists of 9 patients treated with verum and 3 patients treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable patients with left-ventricular dysfunction (LVEF ≤ 45%) after myocardial infarction, whereby the MI occurred 6 or more months before randomization.

  * New York Heart Association (NYHA) class I-II.
  * Left-ventricular ejection fraction ≤ 45%, confirmed by any imaging technique within the last 3 months prior to screening visit will be accepted for screening purposes. If no data are available, an echocardiography has to be performed at screening for inclusion.
  * Treatment with evidence-based therapy for left-ventricular dysfunction post MI for at least 4 weeks prior to screening visit. This therapy has to include at least an Angiotensin-converting enzyme (ACE) inhibitor or an Angiotensin receptor blockers (ARB). Beta-blockers, diuretics, mineralocorticoid receptor antagonist (MRAs), antiplatelet therapy, statins, and aspirin are to be used if indicated. Treatment with stable doses of ACE inhibitors or ARBs using at least half of the recommended target dose (as defined in the European Society of Cardiology (ESC) guidelines, see appendix 16.4) ≥ 4 weeks prior to the screening visit is mandatory.
  * No planned changes to post MI drug therapy during the active treatment phase of the study.
  * Men or confirmed postmenopausal women (defined as being amenorrheic for longer than 2 years with an appropriate clinical profile, e.g. age appropriate and a history of vasomotor symptoms) or women without childbearing potential based on surgical treatment such as bilateral tubal ligation, bilateral oophorectomy or hysterectomy (documented by medical report verification).

Men of reproductive potential must agree to use 2 reliable and acceptable methods for contraception simultaneously when sexually active and not to act as sperm donor. This applies for the time period between signing of the informed consent form and 12 weeks after the last administration of study drug.

Acceptable methods of contraception include, but are not limited to, (i) condoms (male or female) with or without a spermicidal agent; (ii) diaphragm or cervical cap with spermicide; (iii) intra-uterine device; (iv) hormone-based contraception.

* Age: 40 to 79 years (inclusive) at the screening visit.
* Race: Caucasian

Exclusion Criteria:

* Non-ischemic causes for cardiomyopathy will be excluded (including, but not limited to: primary cardiomyopathy, constrictive, restrictive or hypertrophic cardiomyopathy, acute myocarditis, cardiomyopathy secondary to cardiotoxic chemotherapeutic agents).
* Hospitalization for decompensated heart failure within the last 3 months prior to randomization.
* Coronary revascularization within 6 weeks prior to randomization or if revascularization is anticipated or needed during the study duration.
* Clinically relevant, cardiac ischemia in a stress test within 3 months before screening.
* Patients carrying implantable cardioverter defibrillators, cardiac resynchronisation therapy devices or left ventricular assist devices that had any significant clinical events requiring treatment or changes to background medical therapy such as ventricular tachycardias, ventricular fibrillation in the last 6 months before randomization while carrying the devices
* Primary and uncorrected valvular disease with foreseen requirement of valve repair within the next 6 months.
* Any stroke, TIA, any acute coronary syndrome within 6 months prior to randomization.
* Clinically relevant hepatic dysfunction at the screening visit indicated by at least one of the following:
* hepatic insufficiency (Child-Pugh B or C) as documented in medical history
* total bilirubin > 2 times the upper limit normal (ULN) and
* alanine amino transferase (ALT) > 3 times the ULN or
* glutamate dehydrogenase (GLDH) > 3 times the ULN or
* gamma glutamyl transpeptidase (GGT) > 5 times the ULN.
* Systolic blood pressure below 100 or above 160 mm Hg at the screening visit based on the average of 3 readings taken from the arm with the highest recordings.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 20 days
Number of participants with serious adverse events | Up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (10):
- Denmark (4):
  - Copenhagen
  - Copenhagen Ø
  - Hellerup
  - Herlev
- Germany (4):
  - Frankfurt am Main, Hesse
  - Düsseldorf, North Rhine-Westphalia
  - Erfurt, Thuringia
  - Berlin
- Italy (2):
  - Bergamo, Lombardy
  - Brescia, Lombardy